CLINICAL TRIAL: NCT01260090
Title: Vagus Nerve Stimulation to Augment Recovery From Minimally Conscious or Persistently Vegetative States After Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: When Hurricane Sandy hit the area, the funding was pulled.
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Uzma Samadani, Neurosurgeon, VA New York Harbor Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B7301P
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Minimally Conscious States Due to Traumatic Brain Injury; Persistently Vegetative States Due to Traumatic Brain Injury
Keywords: Minimally conscious states; Persistently vegetative states; Traumatic brain injury
MeSH Terms: conditions — Persistent Vegetative State; Brain Injuries, Traumatic | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Vagus Nerve Stimulation (Experimental): Name of the Device:
  We will use the PMA approved version of the NCP System, including the NCP Generator (model 103), NCP Programming Wand (model 201), NCP Programming Software (model 250v7.1), NCP Lead (model 304), NCP Tunneling Tool (model 402) and the Patient Magnet (model 220).
  FDA Facility Registration Number: 1644487
  Interventions: Device: Vagus nerve stimulation;
- No Stimulation (Sham Comparator)
  Interventions: Device: No stimulation

INTERVENTIONS:
Device: Vagus nerve stimulation; — Name of the Device:
  We will use the PMA approved version of the NCP System, including the NCP Generator (model 103), NCP Programming Wand (model 201), NCP Programming Software (model 250v7.1), NCP Lead (model 304), NCP Tunneling Tool (model 402) and the Patient Magnet (model 220).
  FDA Facility Registration Number: 1644487
  Arms: Vagus Nerve Stimulation
Device: No stimulation — Vagus nerve stimulation
  Arms: No Stimulation

SUMMARY:
Traumatic brain injury has a high morbidity and mortality in both civilian and military populations. Blast and other mechanisms of traumatic brain injury damage the brain by causing neurons to disconnect and atrophy. Such traumatic axonal injury can lead to persistently vegetative and minimally conscious states, for which extremely limited treatment options exist, including physical, occupational, speech and cognitive therapies.

More than 50,000 patients have received vagus nerve stimulation for epilepsy and depression. In addition to decreased seizure frequency and severity, patients report enhanced mood, reduced daytime sleepiness independent of seizure control, increased slow wave sleep, and improved cognition, memory, and quality of life.

The purpose of this study is to demonstrate objective improvement in clinical outcome by placement of a vagus nerve stimulator in patients who are recovering from severe traumatic brain injury. Our hypothesis is that stimulation of the vagus nerve results in increased cerebral blood flow and metabolism in the forebrain, thalamus and reticular formation, which promotes arousal and improved consciousness, thereby improving outcome after traumatic brain injury resulting in minimally conscious or persistent vegetative states. If this study demonstrates that vagus nerve stimulation can safely and positively impact outcome, then a larger randomized prospective crossover trial will be proposed.

The investigators will achieve this objective by evaluating whether vagus nerve stimulation impacts clinical recovery from minimally conscious or persistent vegetative states caused by traumatic brain injury as assessed by the FIM™ instrument and Functional Assessment Measure (FIM+FAM) as well as the JFK Coma Recovery Scale Score. The investigators will also evaluate whether vagus nerve stimulation alters resting and activational functional MRI.

Twelve patients will be enrolled in this initial crossover pilot study. These patients will have sustained a severe traumatic brain injury (Disability Rating Scale score of 22 to 29) more than twelve months from starting the study, and have no other concurrent active severe medical problems. Baseline EEG and magnetic resonance imaging (MRI) will be performed prior to left vagus nerve stimulation implantation. Patients will be randomized to alternating three month periods with the device on or off. Outcomes will be assessed at three month intervals with the FIM™ instrument and Functional Assessment Measure (FIM+FAM) and JFK Coma Recovery Scale by a neuropsychologist blinded to the status of the device. Outcomes will also be assessed using quantitative eye movement tracking and functional magnetic resonance imaging. Patients will cross over every 3 months and be followed for at least 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* greater than 12 months from a moderate to severe traumatic brain injury
* Disability Rating Scale score of 18 to 29
* with or without concurrent seizure activity
* Eligible for care in the VA system

Exclusion Criteria:

* Anoxic mechanism of brain injury (eg prolonged arrest)
* Untreated hydrocephalus
* Elevated intracranial pressure
* Systemic issues precluding surgery or 18 months survival
* Traumatic injuries precluding surgery or 18 months survival
* Retained shrapnel or other metal contraindicating MRI
* Prior vagotomy
* Sleep apnea
* Myocardial infarction, arrhythmia
* History of cardiac conduction abnormality
* Pregnancy or intent to become pregnant
* Pre-existing CNS disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
JFK Coma Recovery Scale | every 3 months for 18 months

SECONDARY OUTCOMES:
FIM plus FAM | every 3 months for 18 months
functional MRI | every 3 months for 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Manhattan Va NYHHCS, New York, New York, United States